CLINICAL TRIAL: NCT05130567
Title: A Randomized Study of LP-128 Capsules vs. Placebo to Evaluate Safety, Tolerability and Pharmacokinetics in Healthy Subjects
Brief Title: A Study of LP-128 Capsules in Healthy Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Lupeng Pharmaceutical Company LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP-128-CN101
Record Dates: First submitted 2021-11-09; First posted 2021-11-23 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Single-dose Experimental Group (Experimental): LP-128 capsule will be adminstrated one time at doses up to 240mg
  Interventions: Drug: LP-128 capsules
- Single-dose Control Group (Placebo Comparator): Placebo capsule will be adminstrated one time at doses up to 240mg
  Interventions: Other: Matching Placebo
- Multi-dose Experimental Group (Experimental): LP-128 capsule will be adminstrated once daily, for up to 14 days
  Interventions: Drug: LP-128 capsules
- Multi-dose Control Group (Placebo Comparator): Placebo capsule will be adminstrated once daily, for up to 14 days
  Interventions: Other: Matching Placebo

INTERVENTIONS:
Drug: LP-128 capsules — Oral dosing with LP-128 capsules
  Other Names: NWP-1080
  Arms: Multi-dose Experimental Group; Single-dose Experimental Group
Other: Matching Placebo — Oral dosing with placebo capsules to match LP-128 capsules.
  Arms: Multi-dose Control Group; Single-dose Control Group

SUMMARY:
A Randomized, Double-blind, Placebo-controlled Study to Evaluate Safety, Tolerability and Pharmacokinetics of LP-128 Capsules After Single- and Multiple-Dose in Healthy Subjects

DETAILED DESCRIPTION:
This trial includes single dose and multiple dose phases. The single-dose phase included six dose cohorts. Based on the safety and pharmacokinetic results of single-dose study, approximately 2 doses will be selected to conduct multiple-dose study. The primary study objectives are to evaluate the safety, tolerability, and pharmacokinetic characteristics of LP-128 capsules in healthy subjects after single and multiple dosing.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have no history of serious digestive system, central nervous system, cardiovascular system, kidney, respiratory system, metabolism and endocrine, skeletal and muscular system, blood system disease and cancer
* Subjects (including partners) are willing to take effective contraception measures during study and within 3 months after last dose
* Male and female healthy subjects aged 18 to 55 years old
* Male subjects weigh ≥ 50 kg, and female subjects weigh ≥ 45 kg
* Subjects able to understand and comply with study requirements
* Willing to sign the informed consent and fully understand the content, process and possible adverse reactions of the trial

Exclusion Criteria:

* Abnormal vital signs, physical examination or laboratory tests with clinical significance
* Abnormal ECG, chest X-ray, abdominal ultrasound or echocardiography with clinical significance
* Positive screening for viral hepatitis, HIV and syphilis
* Subjects who have taken any drugs or health care products within 14 or 28 days before administration the study drug; or subjects who have consumed tea or alcohol-containing food product within 24hrs before administration the study drug
* Subjects who have a history of dysphagia or condition may affect drug absorption, distribution, metabolism and excretion
* Female subjects are breastfeeding or pregnant
* Subjects who have a history of drug/alcohol/tobacco abuse
* Subjects who have had a blood donation or massive blood loss within three months before screening; or had major surgery within six months before screening
* Subjects who have participated in other clinical trial within three months before screening
* Subjects have special dietary requirements or cannot tolerate a standard meal
* Subjects who are not suitable for this trial based on the assessment of investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2021-11-19 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) of LP-128 | Up to 4 and 17 days in Single-dose group and Multi-dose group, respectively
  Plasma samples were collected at different points for pharmacokinetic analysis
Apparent terminal phase half-life (T1/2) of LP-128 | Up to 4 and 17 days in Single-dose group and Multi-dose group, respectively
  Plasma samples were collected at different points for pharmacokinetic analysis
Maximum observed plasma concentration (Cmax) of LP-128 | Up to 4 and 17 days in Single-dose group and Multi-dose group, respectively
  Plasma samples were collected at different points for pharmacokinetic analysis
Adverse events of LP-128 | Up to 28 days
  The incidence and severity of adverse events as assessed by NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Excretion of LP-128 in urine | Up to 4 days
  Urine samples will be collected at different points for pharmacokinetic analysis
Excretion of LP-128 in feces | Up to 4 days
  feces samples will be collected at different points for pharmacokinetic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Chongyuan Xu, MD, PhD, Principal Investigator — Nanfang Hospital of Nanfang Medical University
Locations (1):
- NanFang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No